CLINICAL TRIAL: NCT07246213
Title: Improving Cancer Outcomes for Children, Adolescents, and Young Adults: A Multicenter Retrospective Cohort Study on Treatment Failure and Toxicity in Low- and Middle-Income Countries
Brief Title: CAYA Cancer Retrospective Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Resonance, Inc. (Other)
Collaborators: Servier Affaires Médicales (Industry)
Responsible Party: Sponsor
Other Study IDs: RES-NIT-101-25
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-08

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma; Young Adult Cancer; Adolescent Cancer; Childhood Cancers; Acute Lymphoblastic Leukemia (ALL); Lymphoblastic Lymphoma (LBL)
Keywords: Cancer outcomes; Low- and Middle-Income Countries (LMICs); Childhood cancer; Adolescent and young adult cancer (CAYA); Treatment failure; Therapy-related toxicities; Retrospective cohort; Leukemia outcomes; Oncology disparities; High-Income Countries (HICs)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- All Cancer Diagnoses: Patients aged 0-21 years with any type of cancer diagnosis. Retrospective medical record review will capture incidence of treatment failure, including relapse, progression, or abandonment.
  Interventions: Other: Retrospective Medical Record Review
- Acute Lymphoblastic Leukemia / Lymphoblastic Lymphoma: Patients aged 0-21 years diagnosed with acute lymphoblastic leukemia or lymphoblastic lymphoma. Retrospective review will focus on therapy-related toxicities and treatment outcomes in this subgroup.
  Interventions: Other: Retrospective Medical Record Review

INTERVENTIONS:
Other: Retrospective Medical Record Review — This study involves retrospective review of medical records of pediatric, adolescent, and young adult cancer patients (ages 0-21 years) treated at participating oncology centers in Guatemala, Honduras, El Salvador, Armenia, and Tanzania. No experimental drug, device, or behavioral intervention is being administered. Data abstraction will be performed to assess treatment failure, therapy-related toxicities, and clinical outcomes.

SUMMARY:
Despite advances in cancer treatment, significant disparities in outcomes persist between high-income countries (HICs) and low-and middle-income countries (LMICs). Around 80% of children with cancer live in LMICs, where they face challenges such as delayed diagnosis, misdiagnosis, comorbidities, distance to treatment, financial barriers, and limited access to risk-adapted therapies.

Acute lymphoblastic leukemia(ALL)/lymphoblastic lymphoma(LBL), for example, is one of the greatest success stories in pediatric oncology, however, such improvements are not evenly distributed worldwide, and the outcomes for leukemia patients are poorer in LMICs compared to HICs, primarily due to reduced access to quality healthcare.

This study aims to assess cancer treatment outcomes in LMICs, focusing on acute lymphoblastic leukemia/lymphoblastic lymphoma. The findings will inform future studies to implement evidence-based interventions that improve care quality and reduce treatment failures through targeted strategies.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria to be included in this registry:

1. Participants must be willing and able to provide informed consent prior to enrollment in the registry.

   1. For minors or individuals unable to provide informed consent, assent must be obtained along with consent from a legal guardian.
   2. Note: Exemption applies to this criterion when waiver of informed consent/assent is granted by Institutional Review Board(IRB)/Independent Ethics Committee(IEC)/Competent Authorities(CAs).
2. A confirmed diagnosis of any type of cancer within the 15 years prior to the site's activation date.
3. Age 0 to 21 years at the time of diagnosis.
4. Received substantial anti-cancer treatment at the participating center, including but not limited to:

   1. Chemotherapy
   2. Surgery
   3. Radiation therapy
   4. Immunotherapy
5. Medical records are available and accessible for review

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from this registry:

  1. Patients who only visited the participating center for:

     1. Consultation without subsequent primary anti-cancer treatment at the participating center
     2. Pathology, radiology, or other diagnostic evaluations without treatment

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will comprise pediatric patients aged 0-21 years diagnosed with cancer, reflecting diverse demographic backgrounds and clinical characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2028-06-04 (Estimated); Study Completion 2028-12-04 (Estimated)

PRIMARY OUTCOMES:
To estimate the incidence of treatment failure, in patients with any type of cancer diagnosis. | 3 years from date of cancer diagnosis (retrospective follow-up via medical records; patients without an event will be censored at last contact within 3 years)
To estimate the incidence of therapy related toxicities in patients diagnosed with acute lymphoblastic leukemia or lymphoblastic lymphoma. | 3 years from date of cancer diagnosis (retrospective follow-up via medical records; patients without an event will be censored at last contact within 3 years)

SECONDARY OUTCOMES:
To estimate the incidence of treatment failure by cancer type, treatment regimen, age groups, and sociodemographic variables of patients diagnosed with any cancer. | 3 years from date of cancer diagnosis (retrospective follow-up via medical records; patients without an event will be censored at last contact within 3 years)
To estimate the incidence and severity of individual therapy- related toxicities in patients diagnosed with acute lymphoblastic leukemia or lymphoblastic lymphoma. | 3 years from date of cancer diagnosis (retrospective follow-up via medical records; patients without an event will be censored at last contact within 3 years)
To estimate the event-free survival (EFS) and overall survival (OS) for patients diagnosed with acute lymphoblastic leukemia or lymphoblastic lymphoma. | 3 years from date of cancer diagnosis (retrospective follow-up via medical records; patients without an event will be censored at last contact within 3 years)
To describe patterns of relapse in patients with acute lymphoblastic leukemia or lymphoblastic lymphoma. | 3 years from date of cancer diagnosis (retrospective follow-up via medical records; patients without an event will be censored at last contact within 3 years)

CONTACTS AND LOCATIONS:
Locations (5):
- Yeolyan Center for Cancer and Blood Disorders, Yerevan, Armenia
- Fundación Ayúdame a Vivir, El Salvador, El Salvador, El Salvador
- Unidad Nacional de Oncología Pediátrica (UNOP), Guatemala City, Guatemala
- Honduras (2):
  - Hospital Mario Catarino Rivas, San Pedro Sula, Cortés Department
  - Hospital Escuela, Tegucigalpa, Distrito Central

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, the plan for sharing individual participant data (IPD) remains undecided. As the study continues to expand to new sites and additional countries, a comprehensive assessment of applicable data protection and privacy regulations in each jurisdiction is required. A final determination regarding IPD sharing will be made once compliance with all relevant national and international legal frameworks has been ensured.

REFERENCES:
- [Background] Erokhin VV. [Reaction of pulmonary tissue to the administration of weakly virulent Mycobacterium tuberculosis according to histochemical and electron microscopic data]. Arkh Patol. 1969;31(2):19-26. No abstract available. Russian. PMID 4979198
- [Background] Lee TJ, Saito A. Altered cerebral vessel innervation in the spontaneously hypertensive rat. Circ Res. 1984 Sep;55(3):392-403. doi: 10.1161/01.res.55.3.392. PMID 6467529
- [Background] Toft N, Birgens H, Abrahamsson J, Griskevicius L, Hallbook H, Heyman M, Klausen TW, Jonsson OG, Palk K, Pruunsild K, Quist-Paulsen P, Vaitkeviciene G, Vettenranta K, Asberg A, Frandsen TL, Marquart HV, Madsen HO, Noren-Nystrom U, Schmiegelow K. Results of NOPHO ALL2008 treatment for patients aged 1-45 years with acute lymphoblastic leukemia. Leukemia. 2018 Mar;32(3):606-615. doi: 10.1038/leu.2017.265. Epub 2017 Aug 18. PMID 28819280
- [Background] Chantada G, Lam CG, Howard SC. Optimizing outcomes for children with non-Hodgkin lymphoma in low- and middle-income countries by early correct diagnosis, reducing toxic death and preventing abandonment. Br J Haematol. 2019 Jun;185(6):1125-1135. doi: 10.1111/bjh.15785. Epub 2019 Feb 10. PMID 30740656
- [Background] Howard SC, Zaidi A, Cao X, Weil O, Bey P, Patte C, Samudio A, Haddad L, Lam CG, Moreira C, Pereira A, Harif M, Hessissen L, Choudhury S, Fu L, Caniza MA, Lecciones J, Traore F, Ribeiro RC, Gagnepain-Lacheteau A. The My Child Matters programme: effect of public-private partnerships on paediatric cancer care in low-income and middle-income countries. Lancet Oncol. 2018 May;19(5):e252-e266. doi: 10.1016/S1470-2045(18)30123-2. PMID 29726390